CLINICAL TRIAL: NCT02060240
Title: Physical Activity and Obesity: The Role of Nitric Oxide and Eicosanoids in Regulating Capillary Perfusion and Vascular Insulin Resistance
Brief Title: Physical Activity and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Scott M. Chadderdon, Assistant Professor Cardiovascular Medicine, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OHSUIRB#10299; 5KL2TR000152-08 (NIH)
Record Dates: First submitted 2014-02-06; First posted 2014-02-12 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Prediabetic State; Sedentary Lifestyle
Keywords: Obesity; Prediabetic State; Sedentary Lifestyle; Insulin Resistance; Endothelium; Eicosanoids; Nitric Oxide; Regional Blood Flow
MeSH Terms: conditions — Obesity; Prediabetic State; Sedentary Behavior; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Activity Group (Experimental): Subject randomized to High Activity group will have 36, one hour training sessions over 12 weeks.
  Interventions: Behavioral: High Activity
- Standard of Care Group (No Intervention): The standard of care group will maintain their baseline level of activity for 12 weeks

INTERVENTIONS:
Behavioral: High Activity — The high activity group will undergo a 12 week ramped exercise protocol.
  Arms: High Activity Group

SUMMARY:
The purpose of the study is to see if a twelve-week exercise intervention in overweight or obese subjects with pre-diabetes or early disease course type 2 diabetes can lead to improved skeletal muscle capillary blood flow by improving substances that dilate blood vessels and result in improved insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ages 30-60 years of age
2. Overweight and Obese (28< BMI <45)
3. Confirmed pre-diabetic (5.7≤ HbA1c < 6.5)
4. Type 2 DM, Diagnosis 2 years or less, on no medications or metformin only, HbA1c ≤ 6.7

Exclusion Criteria:

1. Stage 3 chronic kidney disease (glomerular filtration rate [GFR] < 60)
2. Obstructive Coronary artery disease
3. Congestive heart failure (ejection fraction < 55%)
4. Peripheral vascular disease,
5. Degenerative joint disease, musculoskeletal disease, or peripheral vascular disease that limits ability to exercise
6. Know hypersensitivity to Definity® ultrasound contrast agent
7. Intra-cardiac or pulmonary shunt
8. The use of antithrombotic agents or a severe bleeding diathesis due to risk of bleeding with intravenous and arterial line placement
9. Physical activity greater than three hours per week
10. Pregnancy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Insulin mediated skeletal muslce blood flow and capillary recruitment | 3 months
  Contrast enhanced ultrasound skeltal muscle perfusion imaging will be performed at rest and during glucose steady state infusion during an insulin clamp. The change in blood flow will be determined between the resting state and at peak steady state to determine the absolute increase in skeletal muslce blood flow (ml/min/g) as well as the absolute increase in capillary blood volume (ml/g) of tissue

SECONDARY OUTCOMES:
Quantification of endothelial derived Vasodilators | 3 months
  To quantify the changes in endothelial derived vasodilators. For this aim nitric oxide bioavailability as tested by flow mediated vasodilation will be performed and reported as absolute change (cm) and percent change (%) in brachial artery diameter from baseline to post ischemic occlusion of the forearm. Plasma samples for eicosanoids will be collected and assessed by liquid chormatography/mass spectroscopy to to assess changes in endothelial derived vasodilators.

OTHER OUTCOMES:
Correalte changes in fitness to vasodilators, blood flow, and insulin sensitivity | 3 months
  Aim 3. To correlate changes in fitness as measured by peak VO2 and anaerobic threshold during cardiopulmonary exercise testing with changes in endothelial derived vasodilators, skeletal muscle blood flow, and insulin sensitivity.

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Chadderdon, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Chadderdon SM, Belcik JT, Smith E, Pranger L, Kievit P, Grove KL, Lindner JR. Activity restriction, impaired capillary function, and the development of insulin resistance in lean primates. Am J Physiol Endocrinol Metab. 2012 Sep 1;303(5):E607-13. doi: 10.1152/ajpendo.00231.2012. Epub 2012 Jun 26. PMID 22739105
- [Background] Coggins M, Lindner J, Rattigan S, Jahn L, Fasy E, Kaul S, Barrett E. Physiologic hyperinsulinemia enhances human skeletal muscle perfusion by capillary recruitment. Diabetes. 2001 Dec;50(12):2682-90. doi: 10.2337/diabetes.50.12.2682. PMID 11723050
- [Background] Clerk LH, Vincent MA, Jahn LA, Liu Z, Lindner JR, Barrett EJ. Obesity blunts insulin-mediated microvascular recruitment in human forearm muscle. Diabetes. 2006 May;55(5):1436-42. doi: 10.2337/db05-1373. PMID 16644702